CLINICAL TRIAL: NCT01299415
Title: A Multi-center, Open-label, Drug-drug Interaction Study to Assess the Effects of Fluvoxamine on the Pharmacokinetics of ASA404 in Adult Patients With Solid Tumor Malignancies
Brief Title: Safety and Pharmacokinetics of ASA404 When Given Together With Fluvoxamine, a Selective Serotonin Receptor Reuptake Inhibitor and CYP1A2 Inhibitor
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASA404A2113
Record Dates: First submitted 2011-01-26; First posted 2011-02-18 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Solid Tumors
Keywords: ASA404,; Phase I,; Oncology,; CYP1A2,; fluvoxamine,; drug drug interaction,; Novartis,; Antisoma
MeSH Terms: conditions — Neoplasms | interventions — vadimezan

ARMS (1):
- ASA404 + Fluvoxamine (Experimental): ASA404 + Fluvoxamine (Core Phase), ASA404 + either paclitaxel or docetaxel or paclitaxel plus carboplain chemotherapy combination (Extension Phase)
  Interventions: Drug: Vadimezan™

INTERVENTIONS:
Drug: Vadimezan™
  Other Names: ASA404

SUMMARY:
This trial is designed to study the drug-drug interaction between ASA404 and fluvoxamine, an inhibitor of its metabolic pathway (CYP1A2). The study will consist of two phases. The purpose of the Core Phase is to study the drug drug interaction between fluvoxamine and ASA404. The purpose of the Extension Phase is to provide continued treatment for those patients that have not progressed during the Core Phase and to collect safety data on ASA404 when given in combination with paclitaxel, docetaxel or the paclitaxel plus carboplatin chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having a histologically-proven and radiologically-confirmed advanced or metastatic solid tumor.
2. WHO Performance Status of 0-2.
3. A minimum of 4 weeks must have elapsed since the last treatment with other cancer therapies.
4. Laboratory values within the ranges, as defined below:

   * ANC ≥ 1.5 X 109 /L
   * Platelets ≥ 100 X 109 /L
   * Hemoglobin ≥ 10 g/dL
   * Serum total bilirubin is within normal range

Exclusion Criteria:

1. Patients having CNS metastasis or evidence of leptomeningeal disease.
2. Patients with any of the following:

   * any clinical or electrocardiographic evidence of cadiac ischemia
   * poorly controlled hypertension
   * family history of unexplained sudden death
   * long QT syndrome
   * history of ventricular fibrillation or torsade de pointes
   * congestive heart failure (NYHA class III or IV)
   * myocardial infarction within 12 months of starting study treatment
3. History of neuroendocrine tumors (e.g. carcinoid tumor, pancreatic islet cell tumor).
4. Significant neurological or psychiatric disorder.
5. Smokers (use of cigarettes within the last 3 months).
6. Concomitant use of drugs that are associated with QTc interval prolongation or have a risk of causing torsade de pointes.
7. Concomitant use of serotonin reuptake inhibitors (SSRIs), 5-hydroxytryptamine (5-HT) receptor agonists or selective serotonin / nor-epinephrine reuptake inhibitors (SNRIs) within 30 days prior to starting study treatment.
8. Concomitant use of somatostain analogues (i.e. octreotide, lanreotide within 30 days prior to starting study treatment.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-08; Primary Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
evaluate the effect of administration of fluvoxamine, a CYP1A2 inhibitor, after 2-cycles of ASA404, on the pharmacokinetics of ASA404 | approximately 2 months

SECONDARY OUTCOMES:
evaluate the effect of administration of fluvoxamine on the safety profile (incidence of AEs or SAEs generated) of ASA404 | 4 months
assess the safety (incidence of AEs and SAEs) of ASA404 in combination with paclitaxel, doctaxel or the paclitaxel plus carboplatin chemotherapy regimen in patients with solid tumor malignancies | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - Univ. of Indiana School of Medicine/Simon Cancer Center, Indianapolis, Indiana
  - Masonic Cancer Center/ Clinical Trials Office, Minneapolis, Minnesota
  - Washington University School of Medicine/Siteman Cancer Center, St Louis, Missouri
  - Cancer Therapy & Research Center, San Antonio, Texas